CLINICAL TRIAL: NCT01338051
Title: The Development of a "Mother/Child, Screen, Treat and Vaccinate Program" in Manchay and Iquitos, Peru (PERCAPS)
Brief Title: The Development of a "Mother/Child, Screen, Treat and Vaccinate Program" in Manchay and Iquitos, Peru
Acronym: PERCAPS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Preventive Oncology International, Inc. (Other)
Collaborators: Peru Instituto Nacional de Enfermadades Neoplasticas (INEN) (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jerome Belinson, Jerome Belinson MD, president, Preventive Oncology International, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PERCAPS I
Record Dates: First submitted 2011-04-16; First posted 2011-04-19 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Cervical Neoplasm; Cervical Dysplasia; Human Papillomavirus
Keywords: Community based participatory research
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Gardasil — Gardasil will be administered to 10-13 year old daughters and granddaughters of study participants according to manufacturers recommended schedule of administration. Gardasil is supplied as 0.5-mL suspension for intramuscular injection at the following schedule: 0, 2 months, 6 months.
  DOSAGE FORMS AND STRENGTHS • 0.5-mL suspension for injection as a single-dose vial and prefilled syringe.

SUMMARY:
This project will use a community based participatory research orientation to develop a model for large scale "campaign" preventive healthcare interventions. The investigators have considerable expertise with cervical cancer screening and HPV vaccination. The investigators also have well tested methodologies for cervical cancer screening that are highly effective, including self-sampling for HPV and improved specimen transport systems. Therefore, the investigators will use these medical interventions as the model preventive health interventions for this project.

DETAILED DESCRIPTION:
Our research group has recently demonstrated that a self-collected cervico-vaginal sample tested with a very high throughput HR-HPV assay is as sensitive has a direct endocervical physician collected sample. Teamed with a non-liquid transport media the investigators believe the technology is solved to reach large populations in a short period of time. With the majority of the world's medically underserved now living in middle income countries it is not necessary to think simple and small to reach the Earth's needy. The investigators can think high tech and high throughput. The massive volumes possible, with proper organization, will control the per/patient cost. The investigators will think "events", not continuous care. Clearly continuous care is the only way to adequately provide the needed care for many problems. However, many interventions can be confined to events which organize large screening or vaccination days and only when positives are identified from the detection algorithm does the healthcare staff become involved for management. The investigators spend an enormous amount of resources identifying the majority of people who will ultimately test negative. The more local the paradigms and the more involved the community in designing the program, the greater will be the participation and the lost to follow-up segment will shrink. This mother, child, screen, treat and vaccinate program will use cervical cancer prevention as the target preventive healthcare intervention. Using community based research orientation the project will begin with a 3 day education program and collaborative meeting with the women leaders of the communities (promotoras). Collectively the investigators will develop the model for the community to advertise, educate, recruit, register, self-collect the specimens, deliver the samples, and report the results. In addition the logistics of the 3 vaccination schedule for the female children will be organized. The medical staff will be involved only with the management of the positives and the vaccine administration. The observational measures will focus on assessing how effectively each of the steps was accomplished.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (adult)

1. Non pregnant women 30-45 years of age in Manchay, and in Iquitos, with female children or grandchildren ages 10-13 who they are willing to enroll in the study to receive Gardasil vaccination.
2. No screening or knowledge of the results of a Pap Test in the last 5 years
3. No hysterectomy
4. No prior pelvic radiation.
5. Willing to sign consent form

Inclusion criteria (children)

1. Female children and grandchildren of a participating women ages 10-13 years
2. No acute illnesses (clinically evident according to vaccinating staff) - such as fever, nausea, vomiting, diarrhea
3. No previous vaccination with Gardasil
4. No reactions to previous dose in their vaccination series
5. No known yeast allergy
6. Willing to participate

Exclusion Criteria:

Exclusion criteria (adults)

Patients will be excluded in the study based on the following criteria:

1. Males
2. Women younger than 30 years old and older than 45 years old.
3. Women without female children or grandchildren age 10-13 or who are unwilling to enroll their 10-13 year old female children or grandchildren to receive Gardasil.
4. Pregnant women.
5. Patients with known history of hysterectomy or radiation for a pelvic cancer.
6. Refusal to participate

Exclusion criteria (Children)

1. Males
2. Girls younger than 10 years old, and older than 13 years.
3. acute illnesses (clinically evident according to vaccinating staff) - such as fever, nausea, vomiting, diarrhea
4. previous vaccination with Gardasil
5. reactions to a previous dose in their vaccination series
6. known yeast allergy
7. Refusal to participate

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 642 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of key study processes used in the process of implementing a mother/child screen, treat and vaccinate program in Iquitos, Peru. | Interview with participants will occur at approximately one month after 2nd vaccination
  The investigators will evaluate community participation, lost to follow up and potential sustainability. One on one interviews with participants will be conducted by trained medical staff. Additional measures to success will be gathered from interviews with promotoras, participating health services staff and recoeded observation. These analyses are descriptive in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome L Belinson, MD, Principal Investigator — Preventive Oncology International; Carlos Vallejos Sologuren, MD, Principal Investigator — Instituto Nacional de Enfermadades Neoplasticas (INEN)
Locations (2):
- Peru (2):
  - Centro de Salud Portada de Manchay, Manchay, Lima region
  - Centro de Salud Bellavista Nanay, Iquitos, Loreto

REFERENCES:
- [Derived] Levinson KL, Abuelo C, Salmeron J, Chyung E, Zou J, Belinson SE, Wang G, Ortiz CS, Vallejos CS, Belinson JL. The Peru Cervical Cancer Prevention Study (PERCAPS): the technology to make screening accessible. Gynecol Oncol. 2013 May;129(2):318-23. doi: 10.1016/j.ygyno.2013.01.026. Epub 2013 Feb 4. PMID 23385153
- See also: Preventive Oncology International — http://www.poiinc.org